CLINICAL TRIAL: NCT07395635
Title: Impact of Immunonutrition in Patients Undergoing Hepatectomies for Liver Tumors: A Randomized Controlled Phase II Trial
Brief Title: Phase II Trial of Immunonutrition in Hepatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Shraddha Patkar, Professor and Surgeon, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study no: 4783
Record Dates: First submitted 2026-01-29; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma; ASA I-III Patients
Keywords: Immunonutrition; Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: Open labelled, Phase II randomized controlled trial Interventional Study
Masking Description: Not Applicable open labelled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Immunomax® Powder- Participant in this group will receive Immunomac Powder 7 consecutive days preceding surgery in a dose of 6-9 scoops (120-180g per day), based on their bodyweight.
  Interventions: Dietary Supplement: Immunonutrition
- Standard Arm (No Intervention): Participant in this group will be advised to continue with their usual oral intake. Patients in this group assessed as having malnutrition will be provided with a standard nutritional supplement (Fortisip®, Nutricia) twice daily (providing 600 kcal energy, 24 g protein), in addition to their usual intake, for the period preceding and including 7 days prior to surgery

INTERVENTIONS:
Dietary Supplement: Immunonutrition — In addition to their usual intake, patients in the intervention arm will be prescribed for each of the 7 consecutive days preceding surgery 6-9 scoops PENTASURE Immunomax® powder (120-180g per day)
  Other Names: PENTASURE IMMUNOMAX POWDER
  Arms: Intervention Arm

SUMMARY:
A randomised open labelled study to evalaute the impact of immunonutrition in Patients Undergoing Hepatectomies for Liver Tumors

DETAILED DESCRIPTION:
Major hepatectomy remains a cornerstone in the curative management of primary and secondary liver tumors. Despite substantial advances in surgical techniques, anesthesia, and perioperative care, hepatectomy continues to be associated with considerable postoperative morbidity and mortality. Reported morbidity rates range from 22% to 40%, while mortality rates vary between 4% and 11%, largely driven by postoperative infectious complications, liver failure, and systemic inflammatory responses. Optimization of preoperative patient status, particularly nutritional and immune function, has therefore emerged as a critical area of interest to improve postoperative outcomes.

Immunonutrition, defined as nutritional supplementation enriched with specific substrates such as arginine, omega-3 fatty acids, and nucleotides, has demonstrated beneficial effects in patients undergoing major gastrointestinal surgery, pancreatic resections, and liver transplantation. These formulations are thought to modulate immune response, attenuate postoperative inflammation, improve protein synthesis, and enhance wound healing. However, evidence supporting the routine use of immunonutrition in patients undergoing hepatectomy remains limited and inconsistent. Existing meta-analyses suggest reductions in postoperative infectious complications and length of hospital stay, but uncertainty persists regarding its overall clinical benefit, particularly in relation to objective nutritional and immunological markers.

The prognostic nutritional index (PNI), calculated using serum albumin levels and total lymphocyte count, is a validated composite marker reflecting both nutritional and immune status. Multiple studies and meta-analyses have shown that a higher preoperative PNI is associated with improved postoperative outcomes and survival following hepatectomy. Furthermore, recent evidence indicates that inflammatory and nutritional biomarkers, including dynamic changes in albumin-based indices, are strong predictors of postoperative morbidity. These findings suggest that targeted immunonutritional interventions capable of improving PNI may translate into meaningful clinical benefits.

Against this background, the present study is designed to evaluate whether preoperative immunonutrition can improve PNI in patients undergoing major hepatectomy for liver tumors. The central hypothesis is that short-term preoperative immunonutrition leads to a measurable improvement in PNI compared with standard nutritional care.

The aim of the study is to assess the effect of preoperative immunonutrition on the prognostic nutritional index in patients planned for major hepatectomy.

The primary objective is to compare the mean change in PNI between patients receiving immunonutrition and those receiving standard nutritional care.

Secondary objectives include evaluating the impact of immunonutrition on postoperative complications, incidence of post-hepatectomy liver failure, length of intensive care unit stay, overall hospital stay, and 90-day postoperative mortality.

This is an open-label, randomized, phase II controlled trial conducted at Tata Memorial Hospital, Mumbai. Adult patients (≥18 years) with liver tumors scheduled for major hepatectomy, defined as resection of three or more liver segments, and classified as ASA physical status I-III will be eligible for inclusion. Patients with severe renal dysfunction, hypersensitivity to immunonutritional components, inability to tolerate oral intake, pregnancy, or conditions impairing informed consent will be excluded.

Eligible patients providing written informed consent will be randomized in a 1:1 ratio into one of two study groups using a centrally generated permuted-block randomization sequence. The intervention group will receive preoperative immunonutrition in addition to their usual oral intake for seven consecutive days prior to surgery. The immunonutritional supplement will be administered in weight-adjusted doses and compliance will be monitored through patient records and telephonic reminders. The control group will continue with their usual oral intake; patients identified as malnourished in this group will receive standard nutritional supplementation as per institutional protocols.

Blood samples will be collected at baseline and repeated on the day prior to surgery to assess serum albumin, lymphocyte count, and inflammatory markers. PNI will be calculated at baseline and preoperatively to evaluate the effect of the intervention. Postoperative assessments will include serial liver function tests, documentation of complications up to 90 days, and recording of ICU and hospital stay durations.

A total of 100 patients (50 per group) will be enrolled over two years, providing adequate power to detect a clinically meaningful difference in PNI between groups. Data will be collected prospectively and analyzed using appropriate statistical methods. Continuous variables will be summarized using means and standard deviations, while categorical variables will be expressed as proportions. The primary endpoint will be analyzed by comparing mean PNI differences between groups, with secondary outcomes evaluated using standard comparative statistical tests.

In summary, this study seeks to generate high-quality prospective evidence on the role of preoperative immunonutrition in improving nutritional and immune status, as measured by PNI, in patients undergoing major hepatectomy. The findings have the potential to inform perioperative nutritional strategies and improve postoperative outcomes in this high-risk surgical population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver tumors planned for major hepatectomies (defined as resection of >/= 3 liver segments)
2. Age above 18 years
3. ASA class I-III

Exclusion Criteria:

1. Preoperative severe renal failure (estimated glomerular filtration rate < 30 ml/min)
2. History of hypersensitivity to arginine, omega-3 fatty acids, or nucleotide 3. Inability to take oral nutrition

4. Pregnancy 5. Mental condition rendering the subject unable to understand the nature, endpoints and consequences of the trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative immunonutrition improves prognostic nutritional index (PNI) | 90 days
  improvement in prognostic nutritional index after maor hepatectomies calculated with the help of Prognostic Nutritional Index (PNI) = [(10 × serum albumin (g/dL)) + (0.005 × total lymphocyte count)].

SECONDARY OUTCOMES:
Incidence of postoperative complications | upto 3 months
  number of complications in both arm major with Clavien-Dindo (CD) classification for adverse events 2. Incidence of post-hepatectomies liver failure (PHLF) 3. Length of ICU stay 4. Length of hospital stay, 5. Incidence of 90 days mortality
Incidence of post-hepatectomies liver failure (PHLF) | Perioperative upto day 5
  nuber of patients undergoing hepatice failure in both study arm after the major hepatectomies define by ndicated by elevated total bilirubin (\(>22\ \mu \text{mol/L}\)) and increased INR (\(>1.2\)) on or after the fifth postoperative day (POD 5), as per ISGLS criteria
Length of ICU stay | Perioperative upto day 30
  number of days participant spent in ICU after hepatectomy till discharge in both treatment group
Length of hospital stay, | Perioperative upto day 30
  number of days participant spent in hospital after hepatectomy till discharge in both treatment group
Incidence of 90 days mortality | Perioperative upto day 90
  death of participant from any cause after the hepatecomy in both treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shraddha Patkar, MD MCh, Principal Investigator — Professor and surgeon
Locations (1):
- Dr. Shraddha Patkar, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang H, Li D, Li J. Prognostic significance of preoperative prognostic nutritional index in hepatocellular carcinoma after curative hepatectomy: a meta-analysis and systemic review. Front Nutr. 2024 Dec 23;11:1433528. doi: 10.3389/fnut.2024.1433528. eCollection 2024. PMID 39764415
- [Result] Solanki SL, Kaur J, Gupta AM, Patkar S, Joshi R, Ambulkar RP, Patil A, Goel M. Cancer related nutritional and inflammatory markers as predictive parameters of immediate postoperative complications and long-term survival after hepatectomies. Surg Oncol. 2021 Jun;37:101526. doi: 10.1016/j.suronc.2021.101526. Epub 2021 Feb 4. PMID 33582497
- [Result] Zhang C, Chen B, Jiao A, Li F, Wang B, Sun N, Zhang J. The benefit of immunonutrition in patients undergoing hepatectomy: a systematic review and meta-analysis. Oncotarget. 2017 Aug 8;8(49):86843-86852. doi: 10.18632/oncotarget.20045. eCollection 2017 Oct 17. PMID 29156839
- [Result] Wong CS, Praseedom R, Liau SS. Perioperative immunonutrition in hepatectomy: A systematic review and meta-analysis. Ann Hepatobiliary Pancreat Surg. 2020 Nov 30;24(4):396-414. doi: 10.14701/ahbps.2020.24.4.396. PMID 33234742
- [Result] Gao B, Luo J, Liu Y, Zhong F, Yang X, Gan Y, Su S, Li B. Clinical Efficacy of Perioperative Immunonutrition Containing Omega-3-Fatty Acids in Patients Undergoing Hepatectomy: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Ann Nutr Metab. 2020;76(6):375-386. doi: 10.1159/000509979. Epub 2020 Dec 11. PMID 33311018
- [Result] Beevi Ss S, Pottakkat B. Effect of Immunonutrition on the Liver Function Status of End-Stage Liver Disease Patients Waiting/Referred for Liver Transplant: A Randomized Controlled Trial. Cureus. 2023 Mar 30;15(3):e36923. doi: 10.7759/cureus.36923. eCollection 2023 Mar. PMID 37128515
- [Result] Zhang G, Zhao B, Deng T, He X, Chen Y, Zhong C, Chen J. Impact of perioperative immunonutrition on postoperative outcomes in pancreaticoduodenectomy: a systematic review and meta-analysis of randomized controlled trials. BMC Gastroenterol. 2024 Nov 16;24(1):412. doi: 10.1186/s12876-024-03510-6. PMID 39550568
- [Result] Markar S, Mariette C, Bonnetain F, Lundell L, Rosati R, de Manzoni G, Bonavina L, Tucker O, Plum P, D'Journo XB, Van Daele D, Cogill G, Santi S, Farran L, Iranzo V, Pera M, Veziant J, Piessen G. Immunonutrition to improve the quality of life of upper gastrointestinal cancer patients undergoing neoadjuvant treatment prior to surgery (NEOIMMUNE): double-blind randomized controlled multicenter clinical trial. Dis Esophagus. 2025 Jan 7;38(1):doae113. doi: 10.1093/dote/doae113. PMID 39863958
- [Result] Franken LC, Schreuder AM, Roos E, van Dieren S, Busch OR, Besselink MG, van Gulik TM. Morbidity and mortality after major liver resection in patients with perihilar cholangiocarcinoma: A systematic review and meta-analysis. Surgery. 2019 May;165(5):918-928. doi: 10.1016/j.surg.2019.01.010. Epub 2019 Mar 11. PMID 30871811
- [Result] van Keulen AM, Buttner S, Erdmann JI, Hagendoorn J, Hoogwater FJH, IJzermans JNM, Neumann UP, Polak WG, De Jonge J, Olthof PB, Koerkamp BG. Major complications and mortality after resection of intrahepatic cholangiocarcinoma: A systematic review and meta-analysis. Surgery. 2023 Apr;173(4):973-982. doi: 10.1016/j.surg.2022.11.027. Epub 2022 Dec 27. PMID 36577599